CLINICAL TRIAL: NCT06046378
Title: The Effect of Digital Stories Prepared With Digital Audio File (Podcast) on Midwifery Learning: A Randomized Controlled Study
Brief Title: The Effect of Digital Stories Prepared With Digital Audio File (Podcast) on Midwifery Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ayla Ergin, Professor Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ayla-1
Record Dates: First submitted 2023-08-10; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Education
Keywords: Digital audio file; podcast; digital story; midwifery; education; natural birth
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Story Group Prepared With Digital Audio File (Podcast) (Active Comparator): The students determined as a result of the randomization will be given a pre-test before the introduction to the "Normal Birth and Postpartum Period " course, which is planned according to the academic calendar. Simultaneously with the subject, digital stories prepared with a digital audio file (podcast) will be sent to the students via e-mail and they will be listened to.
  Interventions: Other: Digital Story Group Prepared With Digital Audio File (Podcast)
- Control (Active Comparator): The students in the control group will listen to the Normal Birth and Postpartum term course face-to-face with the classical education approach. The knowledge level of the students will be measured with the knowledge tests.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Digital Story Group Prepared With Digital Audio File (Podcast) — The students determined as a result of the randomization will be given a pre-test before the introduction to the "Normal Birth and Postpartum Period " course, which is planned according to the academic calendar. Simultaneously with the subject, digital stories prepared with a digital audio file (podcast) will be sent to the students via e-mail and they will be listened to. At the end of the subject on the date planned according to the academic calendar, the students will be interviewed again and a questionnaire will be applied to evaluate the effectiveness of the digital stories prepared with the post-test and digital audio file (podcast). The retention test will be applied 21 days after the last test application.
  Arms: Digital Story Group Prepared With Digital Audio File (Podcast)
Other: Control Group — After the students in the control group are determined, a pre-test will be conducted before the subject receives education. The same knowledge test will be repeated as a post-test after the students receive the classical course education and after the end of the subject. Students will be given a retention test 21 days after the last test. After the retention test application, digital stories prepared with a digital audio file (podcast) will be sent to the students in the control group. In this way, all students participating in the study will have access to the training material used in addition.
  Arms: Control

SUMMARY:
This study was conducted as a randomized controlled study to determine the effect of digital stories prepared with a digital audio file (podcast) on learning in midwifery education. The study was carried out with Kocaeli University Midwifery 3rd grade students. Between October 3 and October 7, 2022, which is the beginning of Kocaeli University 2022-2023 academic year academic calendar, a meeting was held with students about working outside the classroom. The study was completed with 65 students as experimental (n=33) and control group (n=32). Data were collected with participant information form, knowledge test, digital stories evaluation questionnaire prepared with digital audio file (podcast). These stories, which consist of three parts about preparation for natural birth, ideal birth environment and natural birth, were recorded in an appropriate environment and quality, accompanied by a trainer who is an expert in digital audio files (podcast) designs. The knowledge test was applied as a pre-test in the first encounter with the students who accepted the study. Digital stories were sent to the students in the experimental group in the form of e-mails. At the end of the unit, a post-test was administered to both groups. Again, 21 days later, the study was completed by conducting a retention test (knowledge test) and a digital story evaluation questionnaire prepared with a digital audio file (podcast) for both groups. After the study, digital stories prepared with a digital audio file (podcast) were sent to all students in the control group who completed the study, allowing the students to reinforce the subject. While evaluating the findings in the study, Number Cruncher Statistical System 2020 Statistical Software (NCSS LLC, Kaysville, Utah, USA) program was used for statistical analysis. While evaluating the research data, quantitative variables were shown with mean, standard deviation, median, min and max values, and qualitative variables were shown with descriptive statistical methods such as frequency and percentage. Shapiro Wilks test and Box Plot plots were used to evaluate the suitability of the data for normal distribution. Student's t-test, Mann Whitney-U test, Kruskal Wallis test, Dunn test, Spearman correlation analysis, linear regression, chi-square test, Fisher's Exact test, Isher's Exact test and Fisher Freeman Halton and F test were used. The results were evaluated at 95% confidence interval and p<0.05 significance level.

DETAILED DESCRIPTION:
Primary aim: The study is to determine the effect of digital stories prepared with digital audio files (podcasts) on learning in midwifery education.

Hypotheses:

H0: There is no difference between the knowledge test mean scores of the students in the experimental and control groups.

H1: There is a statistically significant difference between the knowledge test mean scores of the experimental and control group students.

H2: There is a statistically significant difference between the satisfaction of the experimental and control group students.

H3: There is no statistically significant difference between the satisfaction of the experimental and control group students.

This study was designed as a randomized controlled experimental study. The study will be carried out at Kocaeli University Faculty of Health Sciences between October 2022-November 2022.

In order to facilitate data collection, the universe of the research will be composed of 70 3rd year midwifery students of Kocaeli University Faculty of Health Sciences in the 2022-2023 academic year. The sample size was based on a study previously published in the literature in 2013 to evaluate the training given to midwifery students on the legal and religious aspects of egg donation through a digital audio file (podcast). The sample calculation was calculated with the G*Power 3.1.9.2 program according to the data of the relevant article.With the obtained values, the effect size was calculated as 0.974. G*Power 3.1.9.2 program effect size and minimum number of students to be included in the study sample: 0.974; a=0.05; power was calculated as 0.95 and the sample size was determined to be less than 16. In order to increase the power of the analysis, the number of samples has been increased and n=16 midwifery students will be included in each group. The experimental group n=16 and the control group n=16) were designed as a digital story prepared in the form of a digital audio file (podcast). In which group the students included in the study will be will be determined from the "Research Lists" website of the random number generation program and will be divided into two groups.

Randomization: The group of mothers will be determined from the random number generator site called "Random Lists". Students will be divided into two groups as experimental and control groups. Thus, the number of each student will be determined and recorded.

Research data were collected by using the Participant Information Form, Knowledge Test and the Questionnaire for Evaluating the Efficiency of Digital Stories Prepared as a Digital Audio File (Podcast).

Exhibitor Information Form: The participant information form was created as a result of the literature review. With this form, students' age, employment status, education status of their parents, the place where they stay during the student period, the place where they provide internet access, the duration and purposes of internet use, the reasons for choosing the midwifery department, the internet usage status in midwifery education and the digital audio file (podcast) before. It includes the situation of listening to the digital story prepared in the form of a digital story and his thoughts on the use of digital stories prepared in the form of a digital audio file (podcast) in midwifery education.

Knowledge test: It was prepared as 50 questions in order to measure the learning levels of the students, the information conveyed by digital stories prepared in the form of digital audio files (podcast). For the knowledge test created, arrangements were made by 10 expert midwife academicians by taking expert opinions. The relevant knowledge test was applied as a pre-test in the first encounter with the students. After listening to the digital stories prepared with a digital audio file (podcast), the experimental group was administered as a post-test and three weeks later as a permanence test.

Digital Stories Prepared with a Digital Audio File (Podcast): The stories created by the researchers as a result of the literature review consisted of three parts: preparation for natural birth, ideal birth environment and storytelling of a natural birth. In the first part, Eda and Melisa's Birth Journey, in the second part, Eda and Melisa's Birth Circle, and in the third part, Eda and Melisa's Meeting Moment. These stories were turned into digital audio files (podcasts) by an educator from Kocaeli University Faculty of Communication who are experts in digital audio files (podcast) designs, in an appropriate environment and quality, and transmitted to the students.

Questionnaire for Evaluating the Efficiency of Digital Stories Prepared with a Digital Audio File (Podcast): It is a form consisting of seven questions and 28 statements and was used to evaluate the effectiveness of digital stories to the experimental group students.

Before the research, a pilot study will be conducted with the 3rd year students of the Department of Midwifery, Faculty of Health Sciences, Selcuk University. This pilot study will be carried out between 26.09.2022 and 30.09.2022 by the researcher using face-to-face interview technique. Students will be asked not to share the study with other students and on social media platforms by signing a consent form and confidentiality agreement.

The main study will be carried out with Kocaeli University Midwifery 3rd year students. Between October 3 and October 7, 2022, which is the beginning of Kocaeli University 2022-2023 academic year academic calendar, a meeting will be held with students about extracurricular work and details will be shared. Participants will be informed that they can leave the research at any time and the study will be completed with volunteer participants. All students participating in the study will sign a confidentiality agreement and it will be ensured that they do not share their work with other students and on platforms such as social media. A participant information form consisting of 22 questions and a knowledge test consisting of 50 statements (pre/post test for natural birth and permanence test) will be applied to both groups.

Randomization will be made among the students who accepted to participate in the study, and two groups will be formed as experimental and control groups. Digital stories prepared with a digital audio file (podcast) will be sent to the students in the experimental group via e-mail. At the end of the relevant topic at the time planned in the academic calendar, a face-to-face interview will be provided to both groups, and a post-test will be applied to both groups. A questionnaire for evaluating the effectiveness of digital stories prepared with a digital audio file (podcast) will be applied to the experimental group students. All students will be given a retention test 21 days after the post-test. After the permanence test is applied, digital stories will be sent to the students in the control group via e-mail.

ELIGIBILITY:
Inclusion Criteria:

* In the 18-30 age range,
* Kocaeli University Faculty of Health Sciences, 3rd year midwifery student,
* Not absenteeism,
* Volunteer to participate in the study and complete the relevant forms,
* No auditory problem,
* Students who have listened to digital audio files (podcasts) at least once
* Able to speak and understand Turkish,
* The mothers who agreed to participate in the study

Exclusion Criteria:

* Those who want to leave the study for any reason during the research process,
* Does not have a mobile phone,
* Have received training on normal birth before,
* Not completing the questionnaires,
* Students who do not listen to digital audio files (podcasts)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Natural birth and non-pharmacological methods information sheet | 1 day (form filled in 30 minutes)
  It will be applied as a pre-test to determine the knowledge level of the students.The knowledge levels of the students about natural birth and non-pharmacological methods were measured. It was prepared as 50 questions by the researchers, each question was evaluated over two points and an evaluation was made out of 100 points. The lowest score of the test is 0, and the highest score is 100. As the score obtained from the test increases, it means that the knowledge level of the students increases. It was administered to all students as a pre-test. Before the Natural Birth and Non-Pharmacological Methods were explained to the students in the Normal Birth and Postpartum Period course.
Natural birth and non-pharmacological methods information sheet | The students in both groups were interviewed it was applied as a post-test 3 weeks after the pre-test (form filled in 30 minutes)
  It will be applied as a post-test to determine the knowledge level of the students.The knowledge levels of the students about natural birth and non-pharmacological methods were measured. It was prepared as 50 questions by the researchers, each question was evaluated over two points and an evaluation was made out of 100 points. The lowest score of the test is 0, and the highest score is 100. As the score obtained from the test increases, it means that the knowledge level of the students increases. It was administered to all students as a pre-test. Before the Natural Birth and Non-Pharmacological Methods were explained to the students in the Normal Birth and Postpartum Period course.
Natural birth and non-pharmacological methods information sheet | The same knowledge test was applied to all students as a retention test 3 weeks after the students took the post-test (Students were given 30 minutes to solve the test)
  The knowledge levels of the students about natural birth and non-drug methods were measured. It was prepared as 50 questions by the researchers, each question was evaluated over two points and an evaluation was made out of 100 points. The lowest score of the test is 0, and the highest score is 100. As the score obtained from the test increases, the knowledge level of the students also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Ergin, Proff. Dr., Principal Investigator — Kocaeli University; Ebru Aktaş, Study Chair — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)